CLINICAL TRIAL: NCT05444868
Title: Validity and Reliability Study of Glittre Activities Of Daily Living Test in Amputees Using Lower Extremity Prosthesis
Brief Title: Validity and Reliability Study of Glittre Activities Of Daily Living Test in Amputees
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Özge Çiftçi, Research Assistant, Eastern Mediterranean University
Other Study IDs: ETK00-2021-0085
Record Dates: First submitted 2022-06-22; First posted 2022-07-06 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Amputation; Traumatic, Limb, Lower
Keywords: Amputees; functional capacity; Glittre ADL; prosthesis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glittre activities of daily living test is used in different populations. The test, which is valid and reliable in different populations, has not been validated in amputees. In our study, we wanted to investigate the validity and reliability of the Glittre activities of daily living test (Glittre ADL) test in amputees using a lower extremity prosthesis.

DETAILED DESCRIPTION:
In individuals with lower extremity amputation, functions such as standing up, sitting, walking, turning, going up and down stairs, going up and down hills, jumping over steps, getting in and out of a car are required. There is no physical function test that simultaneously evaluates both the upper and lower extremities of individuals who have had lower extremity amputations. Therefore, we planned to perform the validity and reliability of the Glittre activities of daily living (ADL) test, which is used in COPD patients, for individuals who have had lower extremity amputation. The Glittre ADL test is the most widely used test to evaluate the performance of COPD patients in activities of daily living. The test is a simple test that can be easily applied and includes functional activities for the lower extremity and upper extremity.

RESEARCH QUESTIONS / HYPOTHESES:

1. Is the Glittre ADL Test reliable in amputees using a lower extremity prosthesis?
2. Is the Glittre ADL Test valid for evaluating amputees using a lower extremity prosthesis?

METHOD OF THE RESEARCH:

Glittre ADL Test:

It is a test that takes place within a distance of 10 m in total. This distance of 10 m will be divided into 2 in the middle by the ladder. Each rung of the ladder will be adjusted 17 cm high and 27 cm deep. Individuals will be asked to climb a 2-step ladder and then walk towards the shelf. The height of the shelves will be adjusted according to the shoulders and waist levels of the participants. It will place 3 pieces of 1 kg objects on the top shelf, one by one, first from the top shelf to the middle shelf, then from the middle shelf to the bottom shelf, from the bottom shelf to the middle shelf, and finally from the middle shelf to the top shelf. It is a test that takes place within a distance of 10 m in total. This distance of 10 m will be divided into 2 in the middle by the ladder. Each rung of the ladder will be adjusted 17 cm high and 27 cm deep. Individuals will be asked to climb a 2-step ladder and then walk towards the shelf. The height of the shelves will be adjusted according to the shoulders and waist levels of the participants. It will place 3 pieces of 1 kg objects on the top shelf, one by one, first from the top shelf to the middle shelf, then from the middle shelf to the bottom shelf, from the bottom shelf to the middle shelf, and finally from the middle shelf to the top shelf.

For the validity test; 2 minute walk test, functional reach test, timed get up and go test will be done and these tests will be examined in terms of Construct validity, Convergent validity and Discriminant validity.

For reliability test; Day 1 and Day 2 will be evaluated by the same physiotherapist. Day 3 will be evaluated by a different physiotherapist.

There will be 3 evaluations in 1 week and it will be planned to be 1 day between evaluations. Two assessments will be done by the same physiotherapist, while the third will be done by another physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* People over the age of 18 who have had lower extremity amputation
* Unilateral amputees using a lower extremity prosthesis for at least 6 months
* Those who can walk at least 30 m independently

Exclusion Criteria:

* Presence of ulcer on the stump
* Lack of stump socket compatibility
* Having a different orthopedic or neurological problem other than amputation
* Having a cardiopulmonary problem that will prevent the test from being completed.
* I ndividuals who cannot understand and follow commands

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Those over the age of 18 who have been using a lower extremity prosthesis for at least 6 months will be included in the study.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Glittre Activities Of Daily Living Test | 3 months
  How long individuals take the Glittre Daily Living Activities Test will be recorded in minutes.

SECONDARY OUTCOMES:
2-Minute Walking Test | 3 months
  The test to be carried out in the 30 meter long area will be marked at 3 meter intervals and the turning points will be determined by an object such as a traffic cone. We will ask the individual to walk the maximum distance in 2 minutes, and we will tell him that he can slow down and stop when he gets tired. When 2 minutes are completed with the stopwatch, we will ask the individual to stop and record the walking distance.
Functional reach test: | 3 months
  The patient will be asked to stand sideways next to the wall and wait with the shoulder flexed at 90 degrees, the elbow extended and the fist closed, without touching the arm close to the wall. The 3rd metacarpal head will be marked and the patient will be asked to lie down as far as he can without stepping, then the new location of the 3rd metacarpal head will be marked. Scoring will be determined by measuring the difference between the start and end position. 3 attempts will be made and the average of the last two trials will be taken.
Timed get up and walk test | 3 months
  The distance of 3 meters in front of the chair will be determined and the individual will be asked to get up from the chair and walk the determined distance.
Trinity Amputation and Prosthetic Experience Scale (TAPES): | 3 months
  TAPES consists of 2 parts. In the first part, psychosocial adaptation, activity limitation and prosthesis satisfaction are questioned, while in the second part, the average number of hours he wears the prosthesis, his physical capacity, general health, stump and phantom pain are questioned. A high score indicates high compliance. A high score in assessing activity limitation indicates activity limitation. Finally, the highest score that can be obtained in the prosthesis satisfaction subscale is 50, the lowest score is 10. A high score indicates that the individual is satisfied with the prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Çiftçi, Bachelor, Principal Investigator — Eastern Mediterranean University; Cansu Koltak, MSc, Principal Investigator — Eastern Mediterranean University; Yasin Yurt, PhD, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Hatfield AG. Beyond the 10-m time: a pilot study of timed walks in lower limb amputees. Clin Rehabil. 2002 Mar;16(2):210-4. doi: 10.1191/0269215502cr484oa. PMID 11911519
- [Background] Mason K, Chockalingam A, Prudhomme S, Stachenko S, Pearson T. Policy depot: a tool to build global capacity in cardiovascular health policy. Glob Heart. 2012 Mar;7(1):47-51. doi: 10.1016/j.gheart.2012.01.005. Epub 2012 Apr 13. No abstract available. PMID 25691167
- [Derived] Ciftci O, Yurt Y, Koltak C, Eker L. Validity and reliability of Glittre activities of daily living test in lower-limb prosthetic users. Prosthet Orthot Int. 2025 Dec 1;49(6):704-709. doi: 10.1097/PXR.0000000000000422. Epub 2024 Dec 24. PMID 39721062
- See also: 2 — http://pubmed.ncbi.nlm.nih.gov/12736892/
- See also: 3 — https://www.semanticscholar.org/paper/Muscle-activation-patterns-during-walking-from-the-Huang-Ferris/2181004661b1d77acbb53523b6071be0aa99f61d
- See also: 4 — http://pubmed.ncbi.nlm.nih.gov/10414769/
- See also: 5 — https://pubmed.ncbi.nlm.nih.gov/11588757/
- See also: 6 — https://pubmed.ncbi.nlm.nih.gov/15982169/
- See also: 9 — https://journals.lww.com/poijournal/Abstract/2012/36040/Selecting_a_test_for_the_clinical_assessment_of.2.aspx
- See also: 11 — https://www.semanticscholar.org/paper/A-field-test-of-functional-status-as-performance-of-Skumlien-Hagelund/b0f8e0121357495498b2fd28e6080ad246184329
- See also: 12 — https://www.semanticscholar.org/paper/Kronik-obstr%C3%BCktif-akci%C4%9Fer-hastalar%C4%B1nda-%C3%A7ok-boyutlu-Kutukcu-Ar%C4%B1kan/709848a1747b1b7d229f6c8a63a028b4486e0e9b